CLINICAL TRIAL: NCT03736213
Title: Correcting Residual Errors With Spectral, Ultrasound, and Traditional Speech Therapy: Delineation of Sensorimotor Subtypes
Brief Title: Delineation of Sensorimotor Subtypes Underlying Residual Speech Errors
Acronym: C-RESULTS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: New York University (Other)
Collaborators: Syracuse University (Other); Montclair State University (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: C-RESULTS-SCED; R01DC017476 (NIH)
Record Dates: First submitted 2018-11-07; First posted 2018-11-09 (Actual); Results first posted 2022-12-29 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2021-12

CONDITIONS: Speech Sound Disorder
Keywords: speech; articulation; motor development
MeSH Terms: conditions — Speech Sound Disorder; Speech

STUDY DESIGN:
Intervention Model Description: In this single-case randomization design, each participant will receive an equal number of sessions of visual-acoustic and ultrasound biofeedback, with randomized allocation of treatment types to individual sessions. Treatment will last 20 hrs (10 days) over a 5 week period. Randomization will be blocked, with each day of treatment serving as a block; within each day, one hour of treatment will be randomly assigned to feature visual-acoustic and one to feature ultrasound treatment. A congruent condition and an incongruent condition will be defined for each participant based on their sensory profile, where the congruent condition is the biofeedback type that is expected to be more effective and the incongruent condition is the type expected to be less effective. Visual-acoustic biofeedback is defined as the congruent condition for individuals with a primary auditory deficit and ultrasound biofeedback is defined as congruent for individuals with a primary somatosensory deficit.
Who Masked: Outcomes Assessor
Masking Description: All perceptual ratings will be obtained from blinded, naive listeners recruited through online crowdsourcing. Following protocols refined in previous published research, binary rating responses will be aggregated over at least 9 unique listeners per token.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Visual-acoustic biofeedback (Experimental): Visual-acoustic biofeedback treatment targeting /r/ distortions.
  Interventions: Behavioral: Visual-acoustic biofeedback
- Ultrasound biofeedback (Experimental): Ultrasound biofeedback treatment targeting /r/ distortions.
  Interventions: Behavioral: Ultrasound biofeedback

INTERVENTIONS:
Behavioral: Visual-acoustic biofeedback — In visual-acoustic biofeedback treatment, the elements of traditional articulatory treatment (i.e., auditory models and verbal descriptions of articulator placement) are enhanced with a dynamic display of the speech signal in the form of the real-time LPC spectrum. Because correct vs incorrect productions of /r/ contrast acoustically in the frequency of the third formant (F3), participants will be cued to make their real-time LPC spectrum match a visual target characterized by a low F3 frequency. I
  Arms: Visual-acoustic biofeedback
Behavioral: Ultrasound biofeedback — In ultrasound biofeedback, the elements of traditional articulatory treatment are enhanced with a real-time ultrasound display of the shape and movements of the tongue. One or two target tongue shapes will be selected for each participant, and a trace of the selected target will be superimposed over the ultrasound screen. Participants will be cued to reshape the tongue to match this target during /r/ production.
  Arms: Ultrasound biofeedback

SUMMARY:
Children with speech sound disorder show diminished accuracy and intelligibility in spoken communication and may thus be perceived as less capable or intelligent than peers, with negative consequences for both socioemotional and socioeconomic outcomes. While most speech errors resolve by the late school-age years, between 2-5% of speakers exhibit residual speech errors (RSE) that persist through adolescence or even adulthood, reflecting about 6 million cases in the US. Both affected children/families and speech-language pathologists (SLPs) have highlighted the critical need for research to identify more effective forms of treatment for children with RSE. In a series of single-case experimental studies, research has found that treatment incorporating technologically enhanced sensory feedback (visual-acoustic biofeedback, ultrasound biofeedback) can improve speech in individuals with RSE who have not responded to previous intervention. Further research is needed to understand heterogeneity across individuals in the magnitude of response to biofeedback treatment.

The overall objective of this proposal is to conduct clinical research that will guide the evidence-based management of RSE while also providing novel insights into the sensorimotor underpinnings of speech. The central hypothesis is that individual deficit profiles will predict relative response to visual-acoustic vs ultrasound biofeedback. From the larger population of children with RSE evaluated as part of C-RESULTS-RCT (Correcting Residual Errors With Spectral, Ultrasound, Traditional Speech Therapy Randomized Controlled Trial), a subset of 8 children will be selected who show a deficit in one domain (auditory or somatosensory) and intact perception in the other. Single-case methods will be used to test the hypothesis that sensory deficit profiles differentially predict response to visual-acoustic vs ultrasound biofeedback.

DETAILED DESCRIPTION:
Single-Case Randomization Component: At the group level, speakers with RSE show poorer auditory and oral somatosensory acuity than typically developing (TD) speakers, but individuals differ in the extent to which each sensory domain is impacted. The objective of this aim is to evaluate how distinct sensory profiles mediate relative response to different types of biofeedback, with the goal of optimizing treatment through personalized learning. This study will test the working hypothesis that visual-acoustic biofeedback will produce larger gains in children whose deficit primarily affects the specification of the auditory target, while ultrasound biofeedback will produce larger gains in children with a primary somatosensory deficit. The main approach to testing this hypothesis is to select, from the larger population of children with RSE evaluated as part of C-RESULTS-RCT, a subset of 8 children who show asymmetric sensory profiles (strong auditory and weak somatosensory acuity, or vice versa). These children will be enrolled in a single-case experimental design where individual treatment sessions are randomly assigned to feature visual-acoustic or ultrasound biofeedback. Participants will complete 20 hrs of treatment (10 days, 2 sessions per day) over a 5 week period. Acoustic measures will be used to evaluate /r/ production accuracy within each session. Randomization tests will be used to evaluate differences in accuracy between ultrasound and visual-acoustic biofeedback treatment conditions.

ELIGIBILITY:
Inclusion Criteria:

* Must be between 9;0 and 15;11 years of age at the time of enrollment.
* Must speak English as the dominant language (i.e., must have begun learning English by age 2, per parent report).
* Must speak a rhotic dialect of English.
* Must pass a pure-tone hearing screening at 20 decibels (dB) Hearing Level (HL).
* Must pass a brief examination of oral structure and function.
* Must exhibit less than thirty percent accuracy, based on trained listener ratings, on a probe list eliciting /r/ in various phonetic contexts at the word level.
* Must show 0-5% accuracy in production of /r/ at the syllable level, based on treating clinicians' perceptual ratings, during an initial Dynamic Assessment phase consisting of 2 hours of traditional (non-biofeedback) instruction.
* Must fit one of two profiles: (1) primary auditory deficit (scores outside the normative predictive interval for auditory measures assessing identification and discrimination of synthetic speech stimuli, but within the normative predictive interval for measures of oral stereognosis and articulator placement awareness or (2) primary somatosensory deficit, with the reverse profile of spared/impaired sensory function.

Exclusion Criteria:

* Must not receive a T score more than 1.3 standard deviations (SD) below the mean on the Wechsler Abbreviated Scale of Intelligence-2 (WASI-2) Matrix Reasoning.
* Must not receive a standard score below 80 on the Core Language Index of the Clinical Evaluation of Language Fundamentals-5 (CELF-5).
* Must not exhibit voice or fluency disorder of a severity judged likely to interfere with the ability to participate in study activities.
* Must not have an existing diagnosis of developmental disability, major neurobehavioral syndrome such as cerebral palsy, Down Syndrome, or Autism Spectrum Disorder, or major neural disorder (e.g., epilepsy, agenesis of the corpus callosum) or insult (e.g., traumatic brain injury, stroke, or tumor resection).
* Must not show clinically significant signs of apraxia of speech or dysarthria.

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Montclair State University, Bloomfield, New Jersey
  - New York University, New York, New York
  - Syracuse University, Syracuse, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Preston JL, McCabe P, Tiede M, Whalen DH. Tongue shapes for rhotics in school-age children with and without residual speech errors. Clin Linguist Phon. 2019;33(4):334-348. doi: 10.1080/02699206.2018.1517190. Epub 2018 Sep 10. PMID 30199271
- [Background] Preston JL, McAllister T, Phillips E, Boyce S, Tiede M, Kim JS, Whalen DH. Treatment for Residual Rhotic Errors With High- and Low-Frequency Ultrasound Visual Feedback: A Single-Case Experimental Design. J Speech Lang Hear Res. 2018 Aug 8;61(8):1875-1892. doi: 10.1044/2018_JSLHR-S-17-0441. PMID 30073249
- [Background] Dugan SH, Silbert N, McAllister T, Preston JL, Sotto C, Boyce SE. Modelling category goodness judgments in children with residual sound errors. Clin Linguist Phon. 2019;33(4):295-315. doi: 10.1080/02699206.2018.1477834. Epub 2018 May 24. PMID 29792525
- [Background] Preston JL, Holliman-Lopez G, Leece MC. Do Participants Report Any Undesired Effects in Ultrasound Speech Therapy? Am J Speech Lang Pathol. 2018 May 3;27(2):813-818. doi: 10.1044/2017_AJSLP-17-0121. PMID 29546269
- [Background] Preston JL, McAllister Byun T, Boyce SE, Hamilton S, Tiede M, Phillips E, Rivera-Campos A, Whalen DH. Ultrasound Images of the Tongue: A Tutorial for Assessment and Remediation of Speech Sound Errors. J Vis Exp. 2017 Jan 3;(119):55123. doi: 10.3791/55123. PMID 28117824
- [Background] Preston JL, Leece MC, Maas E. Motor-based treatment with and without ultrasound feedback for residual speech-sound errors. Int J Lang Commun Disord. 2017 Jan;52(1):80-94. doi: 10.1111/1460-6984.12259. Epub 2016 Jun 14. PMID 27296780
- [Background] Campbell H, Harel D, Hitchcock E, McAllister Byun T. Selecting an acoustic correlate for automated measurement of American English rhotic production in children. Int J Speech Lang Pathol. 2018 Nov;20(6):635-643. doi: 10.1080/17549507.2017.1359334. Epub 2017 Aug 10. PMID 28795872
- [Background] Campbell H, McAllister Byun T. Deriving individualised /r/ targets from the acoustics of children's non-rhotic vowels. Clin Linguist Phon. 2018;32(1):70-87. doi: 10.1080/02699206.2017.1330898. Epub 2017 Jul 13. PMID 28703653
- [Background] McAllister Byun T. Efficacy of Visual-Acoustic Biofeedback Intervention for Residual Rhotic Errors: A Single-Subject Randomization Study. J Speech Lang Hear Res. 2017 May 24;60(5):1175-1193. doi: 10.1044/2016_JSLHR-S-16-0038. PMID 28389677
- [Background] McAllister Byun T, Tiede M. Perception-production relations in later development of American English rhotics. PLoS One. 2017 Feb 16;12(2):e0172022. doi: 10.1371/journal.pone.0172022. eCollection 2017. PMID 28207800
- [Background] McAllister Byun T, Campbell H. Differential Effects of Visual-Acoustic Biofeedback Intervention for Residual Speech Errors. Front Hum Neurosci. 2016 Nov 11;10:567. doi: 10.3389/fnhum.2016.00567. eCollection 2016. PMID 27891084
- [Background] McAllister Byun T, Halpin PF, Szeredi D. Online crowdsourcing for efficient rating of speech: a validation study. J Commun Disord. 2015 Jan-Feb;53:70-83. doi: 10.1016/j.jcomdis.2014.11.003. Epub 2014 Dec 15. PMID 25578293
- [Background] Hitchcock ER, Byun TM, Swartz M, Lazarus R. Efficacy of Electropalatography for Treating Misarticulation of /r/. Am J Speech Lang Pathol. 2017 Nov 8;26(4):1141-1158. doi: 10.1044/2017_AJSLP-16-0122. PMID 28834534
- [Background] Harel D, Hitchcock ER, Szeredi D, Ortiz J, McAllister Byun T. Finding the experts in the crowd: Validity and reliability of crowdsourced measures of children's gradient speech contrasts. Clin Linguist Phon. 2017;31(1):104-117. doi: 10.3109/02699206.2016.1174306. Epub 2016 Jun 7. PMID 27267258
- [Background] Hitchcock ER, Harel D, Byun TM. Social, Emotional, and Academic Impact of Residual Speech Errors in School-Aged Children: A Survey Study. Semin Speech Lang. 2015 Nov;36(4):283-94. doi: 10.1055/s-0035-1562911. Epub 2015 Oct 12. PMID 26458203
- [Background] Hitchcock ER, Byun TM. Enhancing generalisation in biofeedback intervention using the challenge point framework: a case study. Clin Linguist Phon. 2015 Jan;29(1):59-75. doi: 10.3109/02699206.2014.956232. Epub 2014 Sep 12. PMID 25216375
- [Background] Byun TM, Hitchcock ER, Swartz MT. Retroflex versus bunched in treatment for rhotic misarticulation: evidence from ultrasound biofeedback intervention. J Speech Lang Hear Res. 2014 Dec;57(6):2116-30. doi: 10.1044/2014_JSLHR-S-14-0034. PMID 25088034
- [Background] Byun TM, Hitchcock ER. Investigating the use of traditional and spectral biofeedback approaches to intervention for /r/ misarticulation. Am J Speech Lang Pathol. 2012 Aug;21(3):207-21. doi: 10.1044/1058-0360(2012/11-0083). Epub 2012 Mar 21. PMID 22442281
- [Background] Lee S, Potamianos A, Narayanan S. Acoustics of children's speech: developmental changes of temporal and spectral parameters. J Acoust Soc Am. 1999 Mar;105(3):1455-68. doi: 10.1121/1.426686. PMID 10089598
- [Result] Benway NR, Hitchcock ER, McAllister T, Feeny GT, Hill J, Preston JL. Comparing Biofeedback Types for Children With Residual /ɹ/ Errors in American English: A Single-Case Randomization Design. Am J Speech Lang Pathol. 2021 Jul 14;30(4):1819-1845. doi: 10.1044/2021_AJSLP-20-00216. Epub 2021 Jul 7. PMID 34232693

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Institutional review board approval was obtained from the Biomedical Research Alliance of New York (BRANY, protocol number 18-10-393). Participants were recruited via clinical referrals and public notices in the vicinity of the two treatment sites: Syracuse, NY, and Montclair, NJ. Outreach was conducted using recruitment flyers, listserv announcements, and social media posts.
Pre-assignment Details: This study used a within-subjects design. Each participant received both treatment conditions, with sessions randomly assigned to feature one condition or the other.
Units Other Than Participants: Sessions
Groups:
- Visual-acoustic Biofeedback: In visual-acoustic biofeedback treatment, the elements of traditional articulatory treatment (i.e., auditory models and verbal descriptions of articulator placement) are enhanced with a dynamic display of the speech signal in the form of the real-time LPC spectrum. Because correct vs incorrect productions of /r/ contrast acoustically in the frequency of the third formant (F3), participants will be cued to make their real-time LPC spectrum match a visual target characterized by a low F3 frequency.
Period: Overall Study
Arm/Group | Visual-acoustic Biofeedback | Ultrasound Biofeedback
Started | 7; 10 Sessions | 7; 10 Sessions
Completed | 7; 10 Sessions | 7; 10 Sessions
Not Completed | 0; 0 Sessions | 0; 0 Sessions

BASELINE CHARACTERISTICS:
Groups:
- Visual-acoustic Biofeedback and Ultrasound Biofeedback: This study used a within-subjects design. Each participant received two treatment conditions (visual-acoustic biofeedback and ultrasound biofeedback), with sessions randomly assigned to feature one condition or the other.
  Biofeedback--visual-acoustic and ultrasound: In visual-acoustic biofeedback treatment, the elements of traditional articulatory treatment (i.e., auditory models and verbal descriptions of articulator placement) are enhanced with a dynamic display of the speech signal in the form of the real-time LPC spectrum. Because correct vs incorrect productions of /r/ contrast acoustically in the frequency of the third formant (F3), participants will be cued to make their real-time LPC spectrum match a visual target characterized by a low F3 frequency. In ultrasound biofeedback, the elements of traditional articulatory treatment are enhanced with a real-time ultrasound display of the shape and movements of the tongue. One or two target tongue shapes will be selected for each participant, and a trace of the selected target will be superimposed over the ultrasound screen. Participants will be cued to reshape the tongue to match this target during /r/ production.
Arm/Group | Visual-acoustic Biofeedback and Ultrasound Biofeedback
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: months] | 147.1 (32.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Normalized F3-F2 Distance, an Acoustic Measure That Correlates With Perceptual Accuracy of /r/, Measured From /r/ Sounds Produced in Treatment Sessions.
Description: During treatment, one trial in each block of 10 was flagged for measurement and the first three formants (F1, F2, F3) were extracted from the center of the /r/ interval. The distance between the second and third formants (F3-F2) was converted to z-scores relative to normative data from age-matched children with typical speech (Lee et al., 1999). A z-score of 0 represents the mean F3-F2 distance for typical children; a z-score of 1 indicates one standard deviation of the normative sample above the sample mean. Because F3-F2 is small in perceptually accurate /r/, larger values indicate lower accuracy; z-scores above 2 are considered clinically atypical. Summary statistics report the mean and standard deviation of normalized F3-F2 distance for each treatment condition, pooled across participants and sessions. A two-tailed paired-samples t-test (superiority criterion) was used to compare mean normalized F3-F2 distance for each treatment condition across subjects.
Time Frame: Acoustic accuracy was measured in all ten sessions of each type of treatment, which were administered over five weeks.
Population: Note that this study used a within-subjects design. Each participant received both treatment conditions, with individual sessions randomly assigned to feature one condition or the other. Each participant completed 10 sessions of each type.
Measure: Mean (Standard Deviation); unit: Z-score
Groups:
- Visual-acoustic Biofeedback: Visual-acoustic biofeedback: In visual-acoustic biofeedback treatment, the elements of traditional articulatory treatment (i.e., auditory models and verbal descriptions of articulator placement) are enhanced with a dynamic display of the speech signal in the form of the real-time LPC spectrum. Because correct vs incorrect productions of /r/ contrast acoustically in the frequency of the third formant (F3), participants will be cued to make their real-time LPC spectrum match a visual target characterized by a low F3 frequency.
Arm/Group | Visual-acoustic Biofeedback | Ultrasound Biofeedback
Number analyzed (Participants) | 7 | 7
Z-score | 5.73 (6.33) | 6.27 (6.27)
Statistical Analysis 1: Comparison: Visual-acoustic Biofeedback vs Ultrasound Biofeedback; Test type: Superiority; p = .13, paired t-test, two-tailed; df = 6; Mean Difference (Final Values) = .54 — Ultrasound biofeedback treatment condition - visual-acoustic biofeedback treatment condition. Because more accurate productions have lower normalized acoustic values, a negative difference indicates an advantage for US biofeedback

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: The definition of adverse event and serious adverse event used to collect adverse event information does not differ from that of clinicaltrials.gov.
Arm/Group | Visual-acoustic Biofeedback | Ultrasound Biofeedback
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

LIMITATIONS AND CAVEATS:
Single-case randomization designs are limited in that gains from one treatment condition may carry over to the next.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-02-02): https://cdn.clinicaltrials.gov/large-docs/13/NCT03736213/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-02): https://cdn.clinicaltrials.gov/large-docs/13/NCT03736213/SAP_001.pdf